CLINICAL TRIAL: NCT05818943
Title: A Multicenter Study to Assess the Safety, Tolerability, Pharmacokinetics, and Effect on Seizures and Behavioral Symptoms of Multiple Individually Titrated Doses of Radiprodil in Children with GRIN-related Disorder
Brief Title: Honeycomb: Evaluation of Radiprodil in Children with GRIN-related Disorder
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: GRIN Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAD-GRIN-101; 2022-000317-14 (EudraCT Number)
Record Dates: First submitted 2023-02-22; First posted 2023-04-19 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: GRIN-related Disorders
Keywords: GRIN1; GRIN2A; GRIN2B; GRIN2D
MeSH Terms: interventions — radiprodil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Radiprodil (Experimental): Liquid suspension of radiprodil, at concentrations 0.25 mg/mL or 2.50 mg/mL for 1% and 10% formulation respectively. It will be administered twice a day (bid) either orally or via gastric or nasogastric tube, slowly up-titrated to the highest tolerated dose.
  Interventions: Drug: Radiprodil

INTERVENTIONS:
Drug: Radiprodil — Radiprodil is an orally active, negative allosteric modulator of the NR2B subunit of the NMDA receptor.

SUMMARY:
Study RAD-GRIN-101 is a phase 1B trial to assess safety, tolerability, PK, and potential efficacy of radiprodil for the treatment of GRIN-related disorder in children with a Gain-of-Function (GoF) genetic variant. The study is open-label, so all participants will be treated with radiprodil.

Subjects' participation in the study is expected to last up to six months in Part A.

After the end of part A, all participants who are still eligible can choose to continue to receive radiprodil as part of an open-label long-term treatment period (Part B).

DETAILED DESCRIPTION:
The effect of radiprodil is assessed in two (2) cohorts of pediatric participants: one (1) cohort of participants with treatment-resistant seizures (with or without behavioral symptoms) (Cohort 1) and one (1) cohort of participants with behavioral symptoms but no qualifying seizures (Cohort 2) caused by Gain-of-Function (GoF) variants in the GRIN gene. As the daily doses of radiprodil will be individually titrated for every participant and all the participants will receive the study drug, this is in effect a "single group" study.

This study is divided into the following periods:

PART A:

* Screening/Observation Period (35 days): Investigators assess eligibility followed by a four(4)- week Observation Period to evaluate seizure frequency and/or behavioral symptoms.
* Titration Period (approx. 51 days): Overnight stay to administer radiprodil twice daily to assigned dose level, assessing plasma concentrations, safety, and tolerability during the titration period. Once a safe and potentially effective dose has been established, the participant will immediately enter the Maintenance Period.
* Maintenance Period (up to 53 days): During the Maintenance Period, the participant will continue to take the highest safe and potentially effective dose, as identified during the Titration Period. At the end of the Maintenance Period, there will be an additional overnight stay when the participant will either be invited to take part in Part B or enter the Tapering and Safety Follow-up Period.
* Tapering (15 days) and Safety Follow-up Period (14 days): the participant who doesn't take part in the long-term treatment period (Part B) will need to taper off (ie gradually decrease) the study medicine for 15 days and enter a safety Follow-up Period (14 days). In this case, the participant will make one (1) last visit to the study site 14 days after his/her last dose of radiprodil.

PART B:

* Long-Term Treatment Period (not specified): Participation in Part B of the study, at the dose established during part A, will be continued until such time as either the participant withdraws/is withdrawn from the study or sponsor terminates the study. During this period there will be four (4) visits per year, two(2) of which will require overnight stays. At the end of the Long-Term Treatment Period, the participant will enter the Tapering and Safety Follow-up Period.
* Tapering (15 days) and Safety Follow-up Period (14 days): the participant will need to taper off the study medicine for 15 days and enter a safety Follow-up Period of 14 days. In this case, the participant will make one (1) last visit to the study site 14 days after his/her last dose of radiprodil.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥6 months to ≤12 years, with GRIN gene variants known to result in GoF of the NMDA receptor.
* Cohort 1 must have at least 1 observable motor seizure per week and ≥4 observable motor seizures (generalized or focal) during the prospective 4-week Observation Period and must have failed to obtain adequate seizure control with at least 2 antiseizure medications (ASMs) used at appropriate dose and duration.
* Cohort 2 must have significant behavioral and/or motor symptoms based on caregiver report with a CGI-S score ≥4.
* Stable antiseizure therapies and nonpharmacological treatments such as ketogenic diet throughout screening and study participation.

Exclusion Criteria:

* Any other clinically relevant medical, neurologic, or psychiatric condition and/or behavioral disorder unrelated to GRIN-related disorder that would preclude or jeopardize participant's safe participation or the conduct of the study according to the judgement of the investigator.
* Clinically significant laboratory or ECG abnormalities.
* Severe hepatic dysfunction (Child-Pugh grade C).
* History of brain surgery for epilepsy or any other reason.
* Receiving treatment with contraindicated concomitant drugs such as agonists or antagonists of the glutamate receptor, including but not limited to felbamate, memantine, and perampanel.
* Receiving treatment with hormonal therapy such as adrenocorticotrophic hormone or prednisolone.

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2023-03-07 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (TEAEs), Serious TEAEs (SAEs), TEAEs Leading to Discontinuation and Severity of TEAEs | through study completion (average of 2 years).
  Frequency, type, severity and duration of adverse events, serious adverse events and adverse drug reactions.
Maximum Plasma concentration of radiprodil (Cmax) | Titration Visit 1 (week 5): 0,1,2,4,6,8,10,12 hours post-dose. Titration Visits 2,3,4 (week 6 to 11) and Maintenance Visit 4 (week 20): 0,1,2,5 hours post-dose.
Pharmacokinetic plasma concentration of radiprodil: half-life (T1/2) | Titration Visit 1 (week 5): 0,1,2,4,6,8,10,12 hours post-dose. Titration Visits 2,3,4 (week 6 to 11) and Maintenance Visit 4 (week 20): 0,1,2,5 hours post-dose.
Plasma concentration of radiprodil versus time, area under the curve (AUCt) | Titration Visit 1 (week 5): 0,1,2,4,6,8,10,12 hours post-dose. Titration Visits 2,3,4 (week 6 to 11) and Maintenance Visit 4 (week 20): 0,1,2,5 hours post-dose.
Pharmacokinetic plasma concentration of radiprodil, clearance (Cl) | Titration Visit 1 (week 5): 0,1,2,4,6,8,10,12 hours post-dose. Titration Visits 2,3,4 (week 6 to 11) and Maintenance Visit 4 (week 20): 0,1,2,5 hours post-dose.
Pharmacokinetic plasma concentration of radiprodil, Time corresponding to occurrence of Cmax (Tmax) | Titration Visit 1 (week 5): 0,1,2,4,6,8,10,12 hours post-dose. Titration Visits 2,3,4 (week 6 to 11) and Maintenance Visit 4 (week 20): 0,1,2,5 hours post-dose.

SECONDARY OUTCOMES:
Percent change from baseline in V-EEG seizure burden | Baseline (week 5) to study completion (average of 2 years).
  Assessed by 8- to 24- hour video electroencephalogram
Change from baseline in seizure frequency | Baseline (week 5) to study completion (average of 2 years).
  Assessed by seizure diaries
Aberrant Behavior Checklist-Community (ABC-C) | Baseline (week 5) to study completion (average of 2 years).
  The ABCC is a standardized 58-item caregiver-reported problem-behavior rating scale, originally designed to assess treatment effects in people with intellectual disabilities. Each item is scored from 0 (never a problem) to 3 (severe problem). Items load onto one of five empirically derived subscales: Irritability, Agitation, & Crying (15 items); Lethargy/Social Withdrawal (16 items); Stereotypic Behavior (7 items); Hyperactivity/Noncompliance (16 items); and Inappropriate Speech (4 items). A total score would range from 0 to 174.
Caregiver Global Impression of Change (CaGI-C) | Baseline (week 5) to study completion (average of 2 years).
  The CaGI-C is a 7-point caregiver-rated scale ranging from 1 (very much improved) to 7 (very much worse).
Change from Baseline in Clinical Global Impression - Severity [CGI-S] | Baseline (week 5) to study completion (average of 2 years).
  The CGI-S scale is a clinician-rated measures of severity of a symptom or condition, using a single item, 6- or 7-point scale. The CGI-S scale ranges from 1 ("None") to 6 ("Very Severe").
Clinical Global Impression of Change [CGI-C] | Baseline (week 5) to study completion (average of 2 years).
  The CGI scale is a clinician-rated measures of change of a symptom or condition, using a single item, 6- or 7-point scale. The CGI-C scale ranges from 1 ("Very much worse") to 7 ("Very much improved").
Gross Motor Function Measure (GMFM) | Baseline (week 5) to study completion (average of 2 years).
  The GMFM is a standardized observational instrument designed and validated to measure change in gross motor function over time in children with cerebral palsy. There is a 4-point (0 to 3) scoring system for each of the 5 dimensions of gross motor function, with higher scores denoting better performance.
Sleep Disturbance Scale for Children (SDSC) | Baseline (week 5) to study completion (average of 2 years).
  The SDSC is a parent-report measure to screen for sleep disturbances within the preceding period. It is a 27-item questionnaire rated on a 5-point Likert scale, with higher scores being indicative of more acute sleep disturbances.
Pediatric Quality of Life Inventory [PedsQL] | Baseline (week 5) to study completion (average of 2 years).
  The PedsQL is a 23-item generic health status instrument assessing 5 domains of health in children. It's a 0-100 scale, and higher scores are indicative of better health-related quality of life.
Caregiver Burden Inventory (CBI) | Baseline (week 5) to study completion (average of 2 years).
  The CBI is a validated scale providing information regarding the impact of caregiving on the lives of caregivers. It comprises 24 closed questions divided into 5 dimensions. Each dimension includes 4 or 5 items. Each item is given a score between 0 and 4, where higher scores indicate greater caregiver burden.

CONTACTS AND LOCATIONS:
Overall Officials: Vijay Rai, PhD, Study Director — Associate Director of Clinical Operations; Michael Panzara, MD, MPH, Study Chair — Chief Medical Officer
Locations (15):
- United States (2):
  - Mid-Atlantic Epilepsy and Sleep Center, Bethesda, Maryland
  - Columbia University Irving Medical Center, Dept of Neurology, New York, New York
- Queensland Children's Hospital, South Brisbane, Queensland, Australia
- Canada (2):
  - The Hospital for Sick Children (Sick Kids), Toronto, Ontario
  - BC Children's Hospital, Vancouver
- Germany (2):
  - Abteilung für Neuropädiatrie, Klinik und Poliklinik für Kinder - und Jugendmedizin, Universitätsklinikum Leipzig, Leipzig
  - KBO-Kinderzentrum München gemeinnützige GmbH, München
- Italy (2):
  - Istituto di Ricovero e Cura a Carattere Scientifico (IRCCS) - Ospedale Pediatrico Bambino Gesu, Rome, Lazio
  - Azienda Ospedaliero Universitaria Careggi (AOUC) Firenze - Azienda Ospedaliera Universitaria Meyer, Florence, Tuscany
- Netherlands (2):
  - ERASMUS Medisch Centrum, Developmental & Genetic pediatrics, Rotterdam
  - UMC Utrecht - Wilhelmina Kinderziekenhuis, Polikliniek Kinderneurologie, Utrecht
- Spain (2):
  - Universitat de Barcelona - Hospital Sant Joan de Deu Barcelona (HSJDB), Barcelona
  - Hospital Ruber Internacional, Madrid
- United Kingdom (2):
  - Royal Hospital for Children Glasgow, Glasgow
  - Great Ormond Street Hospital For Children NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: Undecided